CLINICAL TRIAL: NCT05849493
Title: Effects and Mechanisms of Change of Internet Delivered Cognitive Behavior Therapy for Generalized Anxiety Disorder Based on Intolerance of Uncertainty or Metacognitive Theory
Brief Title: Effects and Mechanisms of Change of Internet Delivered Cognitive Behavior Therapy for Generalized Anxiety Disorder
Acronym: ORIGAMI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Erik Forsell, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-02380-01-RCT
Record Dates: First submitted 2023-04-04; First posted 2023-05-09 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Generalized Anxiety Disorder
Keywords: internet delivered treatment; digital mental health services; psychiatry; cognitive behavior therapy; intolerance of uncertainty; metacognitive theory; mechanisms of change
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IU-ICBT (Experimental): 10 week program of internet delivered cognitive behavior therapy with written support by licensed clinical psychologist. Based on the Intolerance of uncertainty model of worry.
  Interventions: Behavioral: Intolerance of uncertainty based Internet delivered Cognitive Behavior Therapy
- Meta-ICBT (Experimental): 10 week program of internet delivered cognitive behavior therapy with written support by licensed clinical psychologist. Based on the Metacognitive model of worry.
  Interventions: Behavioral: Metacognitive Internet delivered Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Metacognitive Internet delivered Cognitive Behavior Therapy — Specialist Guided Internet delivered Cognitive Behavior Therapy based on the metacognitive model of excessive worry
  Arms: Meta-ICBT
Behavioral: Intolerance of uncertainty based Internet delivered Cognitive Behavior Therapy — Specialist Guided Internet delivered Cognitive Behavior Therapy based on the Intolerance of uncertainty model of excessive worry
  Arms: IU-ICBT

SUMMARY:
The goal of this clinical trial is to compare two psychological treatments for Generalized Anxiety Disorder. The main questions it aims to answer are:

How well do these treatments work compared to earlier studies? Is one of the treatments more effective than the other? Are the treatments working the way that we think they do? Specifically, do changes in the variables that these treatments aim to target predict changes in anxiety symptoms?

Participants will be randomized to two different internet-based cognitive behavioral therapy (ICBT) programs: Intolerance of uncertainty-based ICBT and metacognition-based ICBT. Both programs consist of 8 treatment modules and run for 10 weeks. A psychologist will respond to the participants assignments and exercises and will respond to messages.

DETAILED DESCRIPTION:
A randomized trial will be conducted within the Internet Psychiatry Clinic in Stockholm. An option will be added to the online sign-up form giving potential patients the option to participate in a treatment for GAD as part of this study. Based on information provided in the sign-up-form and an assessment via video-call with a psychologist, patients will be included/excluded.

Included patients will be randomized (1:1) to two different ICBT treatment programs (IU-ICBT and Meta-ICBT). These programs will be implemented into regular care at the Internet Psychiatry Clinic in Stockholm, meaning that each patient will undergo the regular assessment process at the clinic. Both programs are ICBT programs of similar scope, consisting of 8 modules to be completed during 10 weeks. During this time patients read written material which instructs them to do specific exercises, answer specific questions and can message a psychologist at the clinic via the web-platform. Based on similar treatments on the Internet Psychiatry Clinic we expect around 10% drop-out.

The effectiveness of both forms of ICBT (meaning within-group change in symptoms during the ten-week treatment) will be compared to other ICBT studies on GAD. Our criteria for studies to compare are:

* ICBT as guided self-help, i.e. treatment where the patient is meant to read or otherwise take in pre-written material and is communicating with a psychologist. Not included here are studies on video-call-therapy or chat-bot based treatments.
* Patients are diagnosed with GAD by a professional, either MD or psychologist.
* Either GAD-7 or PSWQ exist as an outcome measure.

When comparing the treatment programs to each other the threshold for a clinically relevant difference will be 3 points on the GAD-7 scale. A simulation based power analysis based on estimates from a pilot study of the IU-ICBT protocol has shown that we have well above 95% power when using mixed models, for that equivalence bound and n = 200 per group. Note however that the parameter estimates that goes into that power-analysis is based on only n = 22 patients. For comparison a more simple power-analysis for a post-treatment t-test show n = 200 gives 95% power (rounded up) for an equivalence bound of d = 0.36. Note that equivalence bounds should normally be justified based on clinical grounds rather than statistical; this latter power analysis is thus for illustrative purposes.

Hypothesis 1: IU-ICBT and Meta-ICBT will be effective and equivalent in a benchmarking analysis. (i.e. the estimated outcome at end of treatment will be equivalent, as defined by our equivalence bounds, and the pre-post change will be comparable to other ICBT studies on GAD).

Data-analysis: We plan to use multi-level modeling to utilize the increased power/precision we get from within-participant repeated measures.

Hypothesis 2: Changes in intolerance of uncertainty will statistically mediate the treatment effect in the IU-ICBT group. Changes in negative metacognitive beliefs about worry will statistically mediate the treatment effect in the Meta-ICBT group. The effect of both mediators will be moderated by level of intolerance uncertainty and negative metacognitive beliefs at baseline. We will also compare the putative mediators to each other with the hypothesis that the mediation-effect will be stronger for the specific mediator that a treatment protocol targets. This last analysis is to be regarded as the most severe test of our mediation analysis.

Data-analysis: Participants will fill out weekly questionnaires which will include our putative mediators (MCQ-30 and IU-12 questionnaires) and their current symptom level (GAD-7 questionnaire). The mediation-effect of both treatment protocols will be analyzed using latent growth curve modeling which is considered suitable for the study of moderation and mediation in clinical trials.

Additional hypotheses: In addition to the primary hypotheses, we may also investigate alternative moderators proposed by the literature. Worry behaviors is hypothesised to moderate treatment effect in the IU-ICBT group since that treatment partially has a behavioral treatment focus. Emotional contrast avoidance will also be investigated as a moderator. We will also explore demographic moderators such as gender and education level.

We will also investigate treatment satisfaction using the client satisfaction questionnaire, and treatment credibility using the treatment credibility scale, as well as patient global impressions of improvement.

ELIGIBILITY:
Inclusion criteria:

* 18 years or older.
* Meet diagnostic criteria for GAD according to DSM-5, as assessed by a psychologist on a video-call.
* Self-rated score > 10 on GAD-7.
* Can read and speak Swedish fluently.
* Have access to a smartphone, tablet, or computer and a Swedish BankID which allows access to the video-calls and treatment platform.
* Have the time and possibility to participate in the 10 week treatment.
* Consents to participate.

Exclusion criteria:

* Patients that are judged to be in greater need of another psychiatric treatment for another psychiatric diagnosis (for example severe depression) and/or is judged to have a high risk of suicide.
* Current drug or alcohol abuse.
* Current severe somatic health concern or social vulnerability if this is judged to be too great an obstacle for the patient to carry out the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-11-27 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Generalized Anxiety Disorder-7 score (GAD-7) | From treatment start to 10 weeks after treatment start
  Measures Generalized Anxiety Symptoms. 7 items. Scores range from 0-21 with higher scores indicating more generalized anxiety
Change in Meta-Cognitions Questionnaire-30 score (MCQ-30, negative meta-cognition sub-scale) | From treatment start to 10 weeks after treatment start
  Putative mediator. The MCQ-30 negative subscale measures negative meta-cognitive beliefs about the danger and uncontrollability of worry. 6 items. Scores range from 6-36 with higher scores indicating more negative beliefs about worry.
Change in Intolerance of Uncertainty Scale-12 score (IUS-12) | From treatment start to 10 weeks after treatment start
  Putative mediator, measures intolerance of uncertainty. 12 items. Scores range from 12-60 with higher scores indicating more intolerance of uncertainty.

SECONDARY OUTCOMES:
Penn-State Worry Questionnaire (PSWQ) | 10 weeks - pre- and post-treatment.
  Measures trait worry. 16 items. Scores range from 16-80 with higher scores indicating more worry.
Contrast Avoidance Questionnaire-Worry (CAQ-W) | 10 weeks - pre- and post-treatment.
  measures Contrast Avoidance related to worry. 25 items. Scores range from 30 to 150 with higher scores indicating a higher degree of using worry to avoid emotional contrasts.
Montomery-Asberg Depression Rating Scale - Self-rated (MADRS-S) | 10 weeks - pre- and post-treatment.
  Measures depression symptoms. 9 items. Scores range from 0 to 54 with higher scores indicating more depressive symptoms.
Meta-Cognitions Qquestionnaire-30 (MCQ-30 - full scale) | 10 weeks - pre- and post-treatment.
  Measures metacognition. 30 items. Scores range from 30-120 with higher scores indicating more potentially dysfunctional metacognitive beliefs about thoughts and worry.
Patient Health Questionnaire-9 (PHQ-9) | 10 weeks - pre- and post-treatment.
  Measures depression symptoms. 9 items. Scores range from 0-27 with higher scores indicating more depressive symptoms.
World Health Organization Disability Assessment Schedule 2.0 | 10 weeks - pre- and post-treatment.
  Measures disability/functional impairment. 12 items. Scores range from 0-48 with higher scores indicating a higher degree of impairment.
Client satisfaction questionnaire (adapted to the clinic) | 10 weeks after treatment start.
  Measures satisfaction with treatment. 8 items. Scores range from 8-32 with higher scores indicating more satisfaction with the treatment.
Worry Behavior Inventory (WBI) | 10 weeks - pre- and post-treatment.
  Inventory of worry behaviors - 10 items. Scores range from 0-40 with higher scores indicating more frequent worry behaviours.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Forsell, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Internet Psychiatry Clinic, Psychiatry Southwest, SLSO, Region Stockholm, Stockholm, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No
Patient records not available to share.